CLINICAL TRIAL: NCT04650217
Title: Combination Treatment With L-DOPA and Exercise for Mood and Mobility Problems in Late-Life
Brief Title: Levodopa and Exercise for Older Adults With Depression and Psychomotor Slowing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated by sponsor (NIMH)
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Bret Rutherford, Associate Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8065; 1K24MH122514-01A1 (NIH)
Record Dates: First submitted 2020-11-17; First posted 2020-12-02 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Depressive Disorder
Keywords: slowed Information processing speed; slowed gait speed
MeSH Terms: conditions — Depressive Disorder | interventions — carbidopa, levodopa drug combination; Exercise; Psychotherapy

STUDY DESIGN:
Intervention Model Description: Double-Blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- L-DOPA + Exercise (Active Comparator): N=20 subjects assigned to L-DOPA + Exercise will receive L-DOPA three times daily for up to 450mg (L-DOPA) and also will receive exercise training 4 times a week (exercise)
  Interventions: Drug: Carbidopa/levodopa; Behavioral: Exercise training
- LDOPA + Control (Active Comparator): N=20 subjects assigned to L-DOPA + Control will receive L-DOPA three times daily for up to 450mg (L-DOPA) and also will receive a stretching and toning regime (Control).
  Interventions: Drug: Carbidopa/levodopa; Behavioral: Control
- Placebo + Exercise (Placebo Comparator): N=20 subjects assigned to Placebo + Exercise will receive placebo three times daily and also will receive exercise training 4 times a week (exercise).
  Interventions: Drug: Placebo; Behavioral: Exercise training
- Placebo + Control (Placebo Comparator): N=20 subjects assigned to Placebo + Control will receive placebo three times daily and also will receive a stretching and toning regime (Control).
  Interventions: Drug: Placebo; Behavioral: Control

INTERVENTIONS:
Drug: Carbidopa/levodopa — L-DOPA is the immediate precursor of dopamine, is converted to dopamine in presynaptic dopaminergic nerve terminals, and enhances dopaminergic transmission in multiple brain regions. Subjects assigned to L-DOPA will begin with a Week 1 L-DOPA daily dosage of 150mg, or 1.5 25mg carbidopa/100mg levodopa tablets at 9am and placebo tablets at
  1pm and 5pm. In Week 2 the L-DOPA daily dose will increase to 300mg (1.5 25mg carbidopa/100mg levodopa tablets at 9am and 5pm, with placebo at 1pm), followed by a Week 3 to 8 L-DOPA daily dose of 450mg (1.5 25mg carbidopa/100mg levodopa tablets three times daily). Subjects assigned to placebo will take 1.5 placebo tablets three times daily for three weeks. Individuals will be instructed to maintain the same timing of doses throughout the study. Individuals unable to tolerate an increased dose will have their dosage reduced to the maximum previously tolerated dose.
  Other Names: sinemet
  Arms: L-DOPA + Exercise; LDOPA + Control
Drug: Placebo — Carbidopa/levodopa matched placebo
  Other Names: Placebo tablet
  Arms: Placebo + Control; Placebo + Exercise
Behavioral: Exercise training — Subjects assigned t Exercise will exercise individually at their home on a program set each week by Dr. Sloan and the research assistant (RA) coach, who will work with the patient to ensure they train according to the program at the appropriate level of intensity. Subjects will select from a series of aerobic activities and for Weeks 1-2 will train at 55-65 percent of maximum HR as established during their qualifying CPET. In Weeks 3-4, they will increase exercise intensity to 65-75 percent of maximum HR, and in Weeks 5-12 they will train at 75 percent of maximum HR.
  Other Names: lifestyle counseling; psychotherapy
  Arms: L-DOPA + Exercise; Placebo + Exercise
Behavioral: Control — Control will engage in a series of stretches and toning exercises designed to promote flexibility and improve core strength.
  Arms: LDOPA + Control; Placebo + Control

SUMMARY:
In this new research study, 80 adults aged > 60 years with a significant depressive disorder and slowed processing and/or gait speed will be randomized to receive levodopa (L-DOPA; which the Candidate has previously shown to increase psychomotor speed and decrease depressive symptoms in older adults), aerobic exercise (itself an effective antidepressant treatment as monotherapy), or their combination in a 2x2 design incorporating placebo and a stretching/toning control. Participants will be evaluated before and after this 12-week duration study across cognitive domains, psychiatric symptoms, gait kinematics and mobility, and task-based magnetic resonance imaging (MRI) focused on effort-based decision making and reward processing. Data from this study will contribute toward the development of improved treatment and prevention strategies to maximize the functioning and active healthspan of older adults with neuropsychiatric disorders.

DETAILED DESCRIPTION:
Late-Life Depression [LLD]), is prevalent, disabling, and associated with high rates of completed suicide. Among the LLD patients at the highest risk of these adverse outcomes are those who manifest decreased processing speed and/or decreased gait speed. To develop urgently needed novel therapeutics for LLD, a reasonable approach is to target systems underlying the development and persistence of psychomotor slowing. One such approach has been to augment dopaminergic signaling since post-mortem experiments and in vivo neuroimaging studies have implicated age-related dopaminergic decline in the development of slowing. L-DOPA is the immediate precursor of dopamine, is converted to dopamine in presynaptic dopaminergic nerve terminals, and enhances dopaminergic transmission in multiple brain regions. As opposed to other dopaminergic interventions (i.e., dopamine receptor agonists and stimulants), a large literature shows beneficial effects of L-DOPA on cognitive performance and gait in patients with Parkinson's disease, all while being a safe and well-tolerated medication that is difficult to differentiate from placebo in terms of side effects.

A second therapeutic strategy that has been tested for LLD and is relevant to psychomotor slowing is aerobic exercise training. A number of reports and meta-analytic reviews suggest that exercise is an effective non-pharmacologic treatment for depression, including depression in older adults. The largest recent study found that progressive aerobic exercise conducted three times weekly for 30min over 24 weeks was effective for depression and was tolerated extremely well (14.3% drop-out rate, 70% intervention adherence). Exercise training may be effective for LLD by counteracting deleterious age-related changes related to its development and maintenance, such as by reducing pro-inflammatory cytokines, normalizing hypothalamic-pituitary-adrenal axis hyperactivity, and decreasing physical disability and social isolation. Exercise also appears to facilitate adaptive neuroplastic changes in the hippocampus, prefrontal cortex (PFC), and anterior cingulate cortex (ACC) as well as increased white matter connectivity.

While both dopaminergic augmentation and exercise are promising interventions, neither treatment alone may be sufficient to address the serious adverse medical and psychiatric outcomes associated with LLD and psychomotor slowing. In our preliminary study (NYSPI IRB# 7270), L-DOPA was associated with significant improvements in gait speed, but the effect size of this improvement was only moderate (d=0.4). L-DOPA failed to increase average gait speed in this study above the 1m/s threshold associated with functional disability and increased mortality risk in epidemiologic samples. While exercise has not been studied specifically in this patient population, meta-analyses of exercise interventions in older adults suggest overall effects on gait speed are modest (d=0.3) and perhaps not clinically significant. Thus, one goal of this study is to combine these interventions having complementary mechanisms of action to realize a greater therapeutic benefit.

This study includes task-based functional MRI that will allow us to probe the differential therapeutic mechanisms of L-DOPA and exercise and further elucidate the nature of effort-based decision making and reward deficits in LLD. Decision making about voluntary behavior requires weighing the benefit of potential rewards against the effort cost required to achieve them. This calculation is performed by separable populations of dopaminergic midbrain neurons whose signals for value and effort are integrated with the ventral striatum (VS). Anterior VS (AVS) consistently has been shown to encode subjective value, increasing with the probability of reward and decreasing with effort discounting, while recent work suggests dorsomedial VS (dmVS) activates during the initiation of effortful action. We hypothesize that older adults are biased toward inactivity (and thereby at risk for depression) on the basis of dopaminergic decline that diminishes subjective value estimates and increases the effort cost of action (i.e., by the development of slowing). Among PD patients, L-DOPA increases willingness to work independently of facilitating movement by increasing subjective value estimates. By increasing fitness and helping individuals learn about their increasing capacities, exercise may facilitate effort initiation. Below, we evaluate whether complementary effects on effortful behavior may be achievable via L-DOPA increasing subjective value and Exercise reducing effort cost.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 60 years
2. Diagnostic and Statistical Manual (DSM) 5 MDD, Dysthymia, or Depression Not Otherwise Specified (NOS)
3. Hamilton Rating Scale for Depression (HRSD) greater than or equal to 18
4. Decreased processing speed (defined as 1 SD below age-adjusted norms on the Digit Symbol Test) or decreased gait speed (defined as average walking speed over 15' course less than 1m/s)
5. Willing to and capable of providing informed consent and complying with study procedures

Exclusion Criteria:

1. Substance abuse or dependence (excluding Tobacco Use Disorder) within the past 12 months
2. History of psychosis, psychotic disorder, mania, or bipolar disorder
3. Probable Alzheimer's Disease, Vascular Dementia, or Parkinson's disease
4. Mini Mental Status Examination (MMSE) less than or equal to 24
5. HRSD suicide item greater than 2 or Clinical Global Impressions (CGI) Severity score of 7 at baseline
6. Current or recent (within the past 4 weeks) treatment with antidepressants, antipsychotics, or mood stabilizers
7. History of allergy, hypersensitivity reaction, or severe intolerance to levodopa/carbidopa
8. Any physical or intellectual disability adversely affecting ability to complete assessments, including physical inability to perform treadmill testing and exercise protocol
9. Acute, severe, or unstable medical or neurological illness
10. Mobility limiting osteoarthritis of any lower extremity joints, symptomatic lumbar spine disease, history of joint replacement surgery, or history of spine surgery
11. Contraindication to magnetic resonance imaging

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret R Rutherford, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 1 participant signed consent to participate, but no one was randomized in the study.
Groups:
- L-DOPA + Exercise; LDOPA + Control; Placebo + Exercise; Placebo + Control: Study terminated, no subjects recruited for this arm.
- Non-randomized Participants: Participants who signed informed consent for the study but were never randomized
Period: Overall Study
Arm/Group | L-DOPA + Exercise | LDOPA + Control | Placebo + Exercise | Placebo + Control | Non-randomized Participants
Started | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant signed consent for the study but was never randomized into a study group
Groups:
- Non-randomized Participants: Participants who signed consent but were not randomized
- Total: Total of all reporting groups
Arm/Group | L-DOPA + Exercise | LDOPA + Control | Placebo + Exercise | Placebo + Control | Non-randomized Participants | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
Age, Customized [Number; unit: years]
  Age |  |  |  |  | 66 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  |  |  | 1 | 1
  Male |  |  |  |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  |  |  | 0 | 0
  Not Hispanic or Latino |  |  |  |  | 1 | 1
  Unknown or Not Reported |  |  |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  |  |  | 0 | 0
  Asian |  |  |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0
  Black or African American |  |  |  |  | 0 | 0
  White |  |  |  |  | 1 | 1
  More than one race |  |  |  |  | 0 | 0
  Unknown or Not Reported |  |  |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: The MADRS is a standard rater-administered measure of depression severity that will be used to measure changes in depressive symptoms during the study.
  The total MADRS score ranges from a minimum score of 0 to a maximum score of 60. Higher scores indicate more severe depression.
Time Frame: Week 0 (Baseline)
Population: 1 participant signed consent to participate in the study but was never randomized to a study group.
Measure: Number; unit: score on a scale
Groups:
- Non-randomized Participants: Participants who consented to participate but were never randomized
Arm/Group | L-DOPA + Exercise | LDOPA + Control | Placebo + Exercise | Placebo + Control | Non-randomized Participants
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
score on a scale |  |  |  |  | 25

ADVERSE EVENTS:
Time Frame: Adverse event data were planned to be collected over the 12 week duration study.
Groups:
- Non-randomized Participants: Participants who consented to participate but were not randomized
Arm/Group | L-DOPA + Exercise | LDOPA + Control | Placebo + Exercise | Placebo + Control | Non-randomized Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04650217/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT04650217/SAP_001.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT04650217/ICF_002.pdf